CLINICAL TRIAL: NCT03716258
Title: Characterizing Biomarkers of Early Parkinson's Disease Progression
Brief Title: Characterizing Biomarkers of Early Parkinson's Disease Progression (TREG)
Acronym: TREG
Status: Terminated | Type: Observational
Why Stopped: COVID-19 Research Restrictions
Sponsor: Oregon Health and Science University (Other)
Collaborators: Portland VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Joseph Quinn, Principle Investigator, Oregon Health and Science University
Other Study IDs: 18545; 4277 (Other: VHAPORHCS)
Record Dates: First submitted 2018-10-20; First posted 2018-10-23 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Parkinson Disease; Movement Disorders
Keywords: Parkinson Disease; Biomarkers; Inflammation
MeSH Terms: conditions — Parkinson Disease; Movement Disorders; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood separated into buffy coat (for T-cells) and optional banking of plasma in a biorepository
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to look at a blood marker of inflammation in early untreated Parkinson's disease.

DETAILED DESCRIPTION:
Objectives:

Parkinson's disease is the second most common neurodegenerative condition worldwide, and while both motor and non-motor symptoms can be improved with symptomatic therapies, there are currently no drugs that slow or halt progression of the disease. All previous trials of neuroprotective therapies have failed, in large part due to the lack of objective, sensitive biomarkers of Parkinson's disease progression.

Plan:

The proposed study aims to characterize the rate of change in a peripheral blood marker of inflammation (Treg percentage) and three quantitative motor measures (finger tapping, 9-hole peg test and peak turn velocity) in a cohort of 25 untreated PD patients with motor testing and blood sampling performed at baseline and at 6 months

Methods:

Participants will have three visits to the Portland VA over a 12 month period. Assessments will be made regarding their Parkinson's disease progression (motor ability and gait and balance). At each visit, a VA phlebotomist will draw whole blood. The VA lab will analyze whole blood for metabolic CBC with differential. The research team will hand carry blood samples from the VA phlebotomist to Dr. Quinn's VA lab in BLDG 103 - E143. A plasma sample will be added to the Neurologic Disorders Repository (MIRB # 3129). Peripheral blood mononuclear cells (PBMC) will be isolated from buffy coats using Ficoll-Paque. The PBMC will be frozen and batch analyzed for T lymphocytes using flow cytometry at OHSU.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 40 and 80 years
* Diagnosis of idiopathic Parkinson's disease based on the UK PD Brain Bank criteria35
* PD diagnosis within 5 years (≤ 5 years)
* Hoehn and Yahr severity stage less than or equal to 3 (Mild to moderate bilateral disease; some postural instability; physically independent).36
* Remain untreated with levodopa or a dopamine agonist for the duration of the study (up to 7 months, can have treatment with MAO-B inhibitors rasagiline or selegiline)
* Able to understand and give informed consent for the study
* Able to stand and walk unassisted

Exclusion Criteria:

* Current use of dopamine-blocking therapy or significant history of dopamine-blocking therapy (> 1 yr of daily use of the following: typical and atypical antipsychotics except for quetiapine and clozapine, metoclopramide, prochlorperazine, tetrabenazine, reserpine)
* Autoimmune disease or current anti-inflammatory or immunomodulatory therapy (aspirin, Tylenol, ibuprofen, naproxen OK)
* Other condition already causing gait dysfunction or likely to cause significant change in motor/gait function over 6 month period (i.e. knee or hip replacement within the past 6 months or surgery planned during the study, peripheral neuropathy causing impaired proprioception at big toes)
* History of treatment with carbidopa/levodopa, dopamine agonist, or amantadine (can have history of treatment with MAO-B inhibitors rasagiline or selegiline)
* Patient anticipates that they will require symptomatic treatment for PD within the next 6 months

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Early, untreated Parkinson's disease
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Peripheral Blood Treg Percentage (1 year) | Enrollment and 12 months
  Change in peripheral blood Treg number (expressed as percentage of total helper T cells) over a 12 month time period in PD patients

SECONDARY OUTCOMES:
Peripheral Blood Treg Percentage (6 months) | Enrollment and 6 months
  Change in peripheral blood Treg number (expressed as percentage of total helper T cells) over a 6 month time period in PD patients

CONTACTS AND LOCATIONS:
Overall Officials: Joseph F Quinn, MD, Principal Investigator — Oregon Health and Science University
Locations (2):
- United States (2):
  - Oregon Health & Science University, Portland, Oregon
  - VA Portland Health Care System, Portland, Oregon

REFERENCES:
- [Result] Monahan AJ, Warren M, Carvey PM. Neuroinflammation and peripheral immune infiltration in Parkinson's disease: an autoimmune hypothesis. Cell Transplant. 2008;17(4):363-72. PMID 18522239
- [Result] Saunders JA, Estes KA, Kosloski LM, Allen HE, Dempsey KM, Torres-Russotto DR, Meza JL, Santamaria PM, Bertoni JM, Murman DL, Ali HH, Standaert DG, Mosley RL, Gendelman HE. CD4+ regulatory and effector/memory T cell subsets profile motor dysfunction in Parkinson's disease. J Neuroimmune Pharmacol. 2012 Dec;7(4):927-38. doi: 10.1007/s11481-012-9402-z. Epub 2012 Oct 11. PMID 23054369
- [Result] Mancini M, Carlson-Kuhta P, Zampieri C, Nutt JG, Chiari L, Horak FB. Postural sway as a marker of progression in Parkinson's disease: a pilot longitudinal study. Gait Posture. 2012 Jul;36(3):471-6. doi: 10.1016/j.gaitpost.2012.04.010. Epub 2012 Jun 29. PMID 22750016
- [Result] Haaxma CA, Bloem BR, Borm GF, Horstink MW. Comparison of a timed motor test battery to the Unified Parkinson's Disease Rating Scale-III in Parkinson's disease. Mov Disord. 2008 Sep 15;23(12):1707-17. doi: 10.1002/mds.22197. PMID 18649395